CLINICAL TRIAL: NCT01521585
Title: A Double-blind, Placebo-controlled Study in Huntington's Disease Patients to Determine the Safety and Tolerability of SEN0014196
Brief Title: A Phase II Safety and Tolerability Study With SEN0014196
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Siena Biotech S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S015-002
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease | interventions — 6-chloro-2,3,4,9-tetrahydro-1H-carbazole-1-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SEN0014196 50 mg oral tablet (Experimental)
  Interventions: Drug: SEN0014196
- SEN0014196 200 mg oral tablet (Experimental)
  Interventions: Drug: SEN0014196
- Placebo tablet (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SEN0014196 — 50 mg oral once daily tablet
  Arms: SEN0014196 50 mg oral tablet
Drug: SEN0014196 — 200 mg oral once daily tablet
  Arms: SEN0014196 200 mg oral tablet
Drug: Placebo — oral once daily tablet
  Arms: Placebo tablet

SUMMARY:
The principal aim of this study is to obtain safety and tolerability data when SEN0014196 is administered orally over 12 weeks to male and female patients with Huntington's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed, manifest HD (CAG repeat length ≥ 36) and motor signs of HD (including motor score of the UHDRS ≥ 5).
* Clinical Stages I to III (Total Functional Capacity Subscale Score [TFC] of ≥ 3).
* Patients must be anticipated to be ambulatory and able to attend outpatient visits for the duration of the study.
* Patients must be aged ≥ 30 years and ≤ 70 years.
* Body mass index between 18 and 31 kg/m2 inclusive, and a body weight greater than 50 kg.
* Patients must be able to give informed consent or have a legal representative who can consent on their behalf. Patients must be able to comply with trial procedures.
* Patients must have no clinically significant and relevant medical or psychiatric history that could affect the conduct of the study and evaluation of the data, as ascertained by the Investigator through detailed medical history and screening assessments.
* Male patients must agree to use condoms during the entire duration of the study and for 3 months following the last dose of study drug.
* Females of childbearing potential (last menses less than 1 year prior to enrolment).

Exclusion Criteria:

* Participation in a study with an investigational drug within 30 days of the Baseline Visit.
* Any prior or concomitant use of Class I or Class II histone deacetylase (HDAC) inhibitors such as Zolinza®/vorinostat or belinostat.
* Clinical evidence of significant or unstable medical illness in the Investigator's judgement, including screening transaminases (AST or ALT) ≥ 3 times the upper limit of normal (ULN), or an estimated GFR < 60 mL/min, or unexplained proteinuria or microscopic haematuria in an uncontaminated sample obtained at Screening and confirmed on repeat testing.
* QTcF interval >450 ms in men and >470 ms in women or PR >220 ms, or other clinically relevant abnormal ECG findings
* Women who are pregnant or breastfeeding.
* Clinically significant abnormalities in the screening laboratory studies which, in the opinion of the Investigator, would interfere with participation in the study.
* Current evidence or history (within 1 year of baseline) of psychosis, hallucinations or delusions, including major depression with psychotic features, as defined in the DSM-IV-TR. Patients currently experiencing mild depression, or moderate depression which is adequately and appropriately treated in the judgment of the Investigator, can participate if depression is not expected to interfere with study participation.
* Suicide risk, as determined by meeting any of the following criteria:

  * A suicide attempt within the past year or suicidal ideation within 60 days of the Baseline Visit (Day 1).
  * Significant risk of suicide, as judged by the Principal Investigator, based on the psychiatric interview or information collected in the C-SSRS.
* Current diagnosis or history (within 1 year of baseline) of any alcohol or substance abuse (except nicotine and caffeine-related disorders) as defined in the DSM-IV-TR.
* Known allergy to any ingredient in the study drug (active and/or placebo).
* A history of malignancy of any type within 2 years prior to screening. A history of surgically excised non-melanoma skin cancers is permitted.
* Any relevant condition, behaviour, laboratory value, or concomitant medication which, in the opinion of the Investigator, makes the patient unsuitable for entry into the study.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2011-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 12 weeks
  Adverse event (AE) reporting, 12-lead electrocardiogram (ECG), vital signs, physical examination findings, and laboratory safety tests. Suicide risk (Columbia Suicide Severity Rating Scale,C-SSRS).

SECONDARY OUTCOMES:
Short-term clinical effects | 12 weeks
  Global Clinical Impression (GCI, patient and clinician-based), UHDRS, Total Motor Scale (UHDRS-TMS), Functional Assessment, Independence Scale Assessment, Problem Behaviours Assessment, Cognitive Battery (Symbol Digit Modalities Test, Stroop Word Test, Verbal fluency, Mini-Mental State Examination [MMSE]).
Modulation of candidate pharmacodynamic markers | 12 weeks
  Acetylation status of mutant huntingtin, levels of soluble huntingtin.
Pharmacokinetic profile | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Reilmann, MD, Principal Investigator — Dept. of Neurology, University of Münster - Germany
Locations (1):
- Dept. of Neurology, University of Münster, Münster, Germany

REFERENCES:
- See also: The European Huntington's Disease Network — http://www.euro-hd.net/html/network